CLINICAL TRIAL: NCT05990660
Title: Bypass Surgery Incorporating a Negative Pressure Renal Assist Device to Resolve AKI
Brief Title: Renal Assist Device (RAD) for Patients With Renal Insufficiency Undergoing Cardiac Surgery
Acronym: BIPASS-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3ive Labs (Industry)
Collaborators: SCIRENT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RAD1117-01
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Renal Insufficiency; Acute Kidney Injury
Keywords: Cardiac Surgery Associated Acute Kidney Injury (CSA-AKI); Renal Compromise; Kidney Disease; Cardiopulmonary Bypass; Renal Assist Device (RAD); Cardiac Surgery
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: BIPASS-AKI is a single-arm, unblinded interventional study designed to assess the safety of the JuxtaFlow System.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: JuxtaFlow System

INTERVENTIONS:
Device: JuxtaFlow System — Mild, controlled negative pressure introduced into the renal pelvis via JuxtaFlow catheters

SUMMARY:
The study is a prospective, non-randomized early feasibility study intended to evaluate the safety and performance of the JuxtaFlow System (also known as the JuxtaFlow Renal Assist Device (RAD)) in participants with pre-existing renal insufficiency who are undergoing cardiac surgery.

DETAILED DESCRIPTION:
The BIPASS-AKI study is intended to evaluate participants who are at an increased risk of developing cardiac surgery-associated acute kidney injury (CSA-AKI), and, subsequently, overall poor outcomes. Patients to be considered for participation include those undergoing elective or urgent in-house on-pump cardiac surgery (to include coronary artery bypass graft, valvular surgery, or combination) and have pre-existing renal insufficiency as defined by a pre-operative eGFR between 15-60 mL/min. Participants meeting inclusion and exclusion criteria will be enrolled into a treatment arm (single-arm study) following the completion of informed consent. Participants will receive implantation of the JuxtaFlow Catheters following completion of the their cardiac surgery while remaining under anesthesia. Treatment with the JuxtaFlow System will be initiated upon the participant's arrival into the intensive care unit and continue for up to 24 hours post-operatively. Preoperative, intra-operative, and post-operative data will be collected on participants to include 15- and 30-day follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate cardiac surgical patients
2. Elective or Urgent on-pump coronary artery bypass grafting (CABG) and/or valvular surgery
3. Age 22 to 85 years
4. eGFR < 60 mL/min/1.73m2
5. Signed informed consent

Exclusion Criteria:

1. End-stage renal disease (receiving hemodialysis or glomerular filtration rate <15 ml/min/1.73m2)
2. Planned off-pump surgery
3. Any patients with high-grade proteinuria (i.e., urine protein concentration > 300 mg/dL)
4. Pregnancy
5. Any secondary condition as determined by the investigator that would place the subject at an increased risk, or preclude the subject's full compliance with the study procedures, including injuries to the urinary organs and/or external genitals
6. Current or planned treatment with an investigational drug (IND), device (IDE), or other investigational intervention within 3 months prior to or during participation in this clinical trial

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
[Safety] Adverse Events Characterization | 30 days
  The characterization of all type, frequency, severity, and device-relatedness of the adverse events (AEs) associated with the placement, use, and removal of the JuxtaFlow System for the treatment of renal insufficiency in cardiac surgery patients.
[Efficacy] Creatinine Clearance | 24 hours
  The change in measured creatinine clearance occurring over the treatment period of 24 hours or less.
[Efficacy] Urine Sodium Excretion | 24 hours
  The change in urine sodium excretion occurring over the treatment period of 24 hours or less.

CONTACTS AND LOCATIONS:
Overall Officials: Slobodan Micovic, MD, Principal Investigator — Institute for Cardiovascular Diseases Dedinje; Milovan Petrovic, MD, Principal Investigator — Institute of Cardiovascular Diseases of Vojvodina
Locations (3):
- Polsko-Amerykanskie Kliniki Serca, Centrum Kardiologii, Krakow, Bielsko-Biata, Poland
- Serbia (2):
  - Institute for Cardiovascular Diseases "Dedinje", Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz

IPD SHARING:
Plan to Share IPD: No